CLINICAL TRIAL: NCT03647436
Title: Prospective Cohort Study on the Incidence of Geriatric Syndromes Overlap in Patients With Hospital Admission Due to Hip Fracture
Brief Title: Incidence of Geriatric Syndromes Overlap
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital de la Ribera (Other)
Responsible Party: Principal Investigator, Francisco Jose Tarazona-Santabalbina, Principal Investigator, Hospital de la Ribera
Other Study IDs: HULRCP31072018
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: GERIATRIC SYNDROMES; Hip Fractures; GERIATRIC ASSESSMENT; Delirium; Depression; Malnutrition
MeSH Terms: conditions — Hip Fractures; Delirium; Depression; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Elderly patients with hospital admission due to hip fracture and score less than 12 points in the short-MNA at the moment of hospital admission.
  Intervention:
  Comprehensive Geriatric Assesment (CGA). Both groups.
  CGA includes measuring of:
  Previous functional assessment of daily life activities (Barthel and Lawton index), a cognitive screening (MiniMental State Examination), the turn-based assessment of the presence of delirium (Confusion Assessment Method) and in case of presence of delirium will be measured the duration and intensity of the symptoms (Delirium Rating Scale-Revised-98). Likewise, the presence of frailty (Clinical Frailty Scale) and walking ability (Functional Ambulation Categories) will be evaluated.
  Interventions: Other: Comprehensive Geriatric Assessment. Both groups.
- Control group: Elderly patients with hospital admission due to hip fracture and score equal or higher than 12 points in the short MNA at the moment of hospital admission
  Intervention:
  Comprehensive Geriatric Assesment (CGA). Both groups.
  CGA includes measuring of:
  Previous functional assessment of daily life activities (Barthel and Lawton index), a cognitive screening (MiniMental State Examination), the turn-based assessment of the presence of delirium (Confusion Assessment Method) and in case of presence of delirium will be measured the duration and intensity of the symptoms (Delirium Rating Scale-Revised-98). Likewise, the presence of frailty (Clinical Frailty Scale) and walking ability (Functional Ambulation Categories) will be evaluated.
  Interventions: Other: Comprehensive Geriatric Assessment. Both groups.

INTERVENTIONS:
Other: Comprehensive Geriatric Assessment. Both groups. — Evaluation of the incidence of geriatric syndromes: depression, delirium, cognitive disorders, falls, gait disturbances, urinary and fecal incontinence

SUMMARY:
The overlap of depression and delirium as geriatric syndromes present in elderly patients with hospital admission due to hip fracture has been previously studied. Nevertheless, the relationships between these two clinical processes and other geriatric syndromes, especially malnutrition, have not been studied. For this reason, a prospective cohort study has been designed to know the differences in the incidence of geriatric syndromes during hospital admission due to hip fracture in patients with and without risk of malnutrition.

DETAILED DESCRIPTION:
The hypothesis of this work is that in patients with malnutrition, the incidence of overlap between delirium and depression is higher and causes worse health outcomes during hospital admission due to hip fracture. In addition, an increase in the incidence of other geriatricBoth groups. syndromes could be observed, increasing the severity of the known overlap.

Methods:

Objectives:

Main outcome: To evaluate the increase in the incidence of overlap between delirium and depression in patients with malnutrition with respect to patients without malnutrition and to check their influence on quality of care management indicators in patients admitted for hip fracture.

Secondary outcomes:

To estimate the difference in in-hospital mortality and at 12 months between both groups.

To estimate the influence of the joint incidence of the three geriatric syndromes on:

* Number of hospital complications.
* Hospital stay
* Functional recovery.

Type of study:

A cohort study has been designed. Study period: August 2018- December 2019. Scope: Patients aged ≥70 years admitted to the University Hospital of La Ribera (HULR) with the main diagnosis of hip fracture (ICD 9 820.**).

Eligibility criteria Inclusion criteria Patients ≥70 years admitted to the University Hospital of La Ribera (HULR) with the main diagnosis of hip fracture (ICD 9 820.**) undergoing surgery.

Exclusion criteria Life expectancy less than 3 months Dementia GDS 7 that prevents collaboration in the completion of the scale of Global Depression of Yesavage.

Sample size:

Considering a hospital mortality of 11% in patients with delirium, compared to 4% obtained in the total of patients hospitalized for hip fracture in the period 2012-2016 in the HULR with an alpha error of 5% and a beta error of 15 % the sample size is 253 patients per group. The power of the study is 98.5%.

Study variables:

Age Gender Birthdate Date of admission Date of intervention Charlson Index Barthel scale for basic activities of daily life (Prior to admission, admission and discharge) Yesavage Depression Scale (15 items) Short-MiniNutritional Assessment (MNA) Scale Confusion Assessment Method (CAM) delirium Delirium Rating Scale-Revised-98 (DRS-R-98) scale of delirium intensity. Functional Ambulation Categories (FAC) walking scale Hospital mortality 365-day mortality Analytical parameters: Total cholesterol mg / dl Total protein g / dl Albumin g / dl Lymphocytes 109mm3 Calcidiol ng / ml Parathormone (PTH) μg / ml

Follow-up Survival and ambulatory capacity will be monitored 365 days after hospital discharge through access to the electronic medical record.

Statistic analysis The data will be analyzed with the statistical software program Statistical Package for the Social Sciences (SPSS) version 22 (SPSS Inc., Chicago, IL).

A description of the qualitative variables (including dichotomous) will be made by using absolute and relative frequencies. For the quantitative variables, measures of central tendency (mean and median), measures of position (median and quartiles next to box and whisker diagram), dispersion measures (range, interquartile range, variance and standard deviation) and measures of kurtosis will be used. and asymmetry.

The baseline differences between the groups will be analyzed by pruebas2 tests for categorical variables, using Fisher's exact test when any of the expected frequencies does not reach 5 units.

For the variables of quantitative type, with normality verified by the Kolmogorov-Smirnov test, to compare means between the different groups, we will use the T test for independent samples, in the dichotomous variables, and by means of ANOVA of a factor, in the variables with three or more categories. Non-parametric tests will be used: Mann-Whitney U, for dichotomous variables and Kruskal-Wallis for variables with three or more categories otherwise. Multiple comparisons between groups were analyzed using the Bonferroni test in the case of homoscedasticity and by the Games-Howell test in the case of heteroskedasticity, analyzed by the Levene's test.

For the analysis of the main objective, a survival analysis will be carried out using the Kaplan-Meier technique. Likewise, the Hazard Ratio of the mortality risk will be calculated by means of a Cox regression, using as confusing variables those considered as such in the analysis of the functioning of the randomization and those that, in the opinion of the investigators, present relevant clinical importance.

Finally, the calculation of the relative risks (RR) will be carried out together with its confidence interval at 95% of the incidence of hospitalizations and the ability to wander. A survival analysis will be performed using the Kaplan-Meier technique for each variable related to the secondary objectives. A Cox regression will be performed for each variable of the secondary objectives, using as confusing variables those considered as such in the analysis of the functioning of the randomization and those that, in the opinion of the researchers, present relevant clinical importance.

Limitations Those derived from a non-randomized study. To avoid interobserver variability, a trainer will be made with the personnel in charge of administering the scales together with a brief pilot study in which the agreement will be analyzed using the Kappa statistical test.

ELIGIBILITY:
Inclusion Criteria:

Patients ≥70 years admitted to the University Hospital of La Ribera (HULR) with the main diagnosis of hip fracture (ICD 9 820. **) that are going to be operated on.

Exclusion Criteria:

Life expectancy less than 3 months Dementia GDS 7 that prevents collaboration in the completion of the scale of Global Depression of Yesavage.

Min Age: 70 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients aged ≥70 years admitted to the University Hospital of La Ribera (HULR) with the main diagnosis of hip fracture (ICD 9 820. **).
Sampling Method: Non-Probability Sample
Enrollment: 506 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression and delirium overlap | "4 weeks"
  To evaluate the incidence of overlap between delirium and depression in patients with malnutrition compared to patients without malnutrition
  Measures:
  Prevalence of depression in admitted patients using Geriatric Depression Scale (GDS) of Yesavage. 15-items version. Range 0 to 15 points. Depression is considered with 7 or more points.
  Incidence of depression in admitted patients using Confusion Assessment Method (CAM). Range 0 to 4 points. CAM is considered positive for delirium with 3 points.

SECONDARY OUTCOMES:
Hospital complications | "4 weeks"
  To estimate :
  - Number of hospital complications (surgical wound infection, pneumonia, pressure sores, urinary tract infection, sepsis, Deep Venous Thrombosis, Pulmonary embolism)
Hospital length of stay (days) | "4 weeks"
  Measured in days
Functional recovery. | "4 weeks"
  Functional Ambulation Categories scale (FAC). Range 0 to 5. Positive functional recovery 2 or more points.
  Barthel Index for Activities of Daily Living. Range 0 to 100. <20 points: total dependence. 20-35 points: severe dependence. 40-55 points: moderate dependence.
  ≥ 60 points: mild dependence. 100 points: independence. The Lawton Instrumental Activities of Daily Living Scale. Range 0 to 8 Instrumental dependency 4 points or lower score
Survival | "1 year"
  To estimate the difference in in-hospital mortality and at 12 months between both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Tarazona-Santabalbina, MD, PhD, Principal Investigator — Hospital Universitario de la Ribera
Locations (1):
- Hospital Universitario de la Ribera, Alzira, Kingdom of Valéncia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Downing LJ, Caprio TV, Lyness JM. Geriatric psychiatry review: differential diagnosis and treatment of the 3 D's - delirium, dementia, and depression. Curr Psychiatry Rep. 2013 Jun;15(6):365. doi: 10.1007/s11920-013-0365-4. PMID 23636988
- [Background] Radinovic KS, Markovic-Denic L, Dubljanin-Raspopovic E, Marinkovic J, Jovanovic LB, Bumbasirevic V. Effect of the overlap syndrome of depressive symptoms and delirium on outcomes in elderly adults with hip fracture: a prospective cohort study. J Am Geriatr Soc. 2014 Sep;62(9):1640-8. doi: 10.1111/jgs.12992. PMID 25243678